CLINICAL TRIAL: NCT01524016
Title: 68Ga-DOTATATE PET/CT for Detection and Evaluation of the Causative Tumor of Oncogenic Osteomalacia
Brief Title: 68Ga-DOTATATE PET/CT in Oncogenic Osteomalacia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM001
Record Dates: First submitted 2012-01-29; First posted 2012-02-01 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2014-07

CONDITIONS: Oncogenic Osteomalacia; Mesenchymal Tumor
Keywords: Oncogenic osteomalacia; mesenchymal tumor; Somatostatin receptor; 68Ga-DOTATATE; PET/CT
MeSH Terms: conditions — Oncogenic osteomalacia | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-DOTATATE, PET/CT scan (Experimental): We will perform 68Ga-DOTATATE PET/CT scanning on subjects
  Interventions: Drug: 68Ga-DOTATATE

INTERVENTIONS:
Drug: 68Ga-DOTATATE — Intravenous injection of one dosage of 72-185MBq (2-5 mCi) 68Ga-DOTATATE solution. Tracer doses of 68Ga-DOTATATE will be used to image tumors by Positron Emission Tomography / computed tomography (PET/CT)
  Other Names: (68)Ga-DOTA-d-Phe(1),Tyr(3)-octreotate

SUMMARY:
Oncogenic osteomalacia is rare disease predominantly caused by a small, somatostatin receptor positive mesenchymal tumor, which is frequently hidden in an unusual anatomical site and often goes undetected by conventional imaging. A permanent cure of the disease relies on exactly localizing the tumor and completely removing it. 68Ga-DOTATATE PET/CT is a novel scan that might have improved sensitivity and resolution specifically for somatostatin receptor positive tumors. The investigators will scan the suspicious and confirmed patients of oncogenic osteomalacia and compare it to 99mTc-HYNIC-TOC SPECT/CT and 18F-FDG PET/CT to see if it improves patient care.

DETAILED DESCRIPTION:
Oncogenic osteomalacia, or tumor-induced osteomalacia, is a rare, serious paraneoplastic syndrome. It is predominantly driven by a small, benign mesenchymal tumor. The disease is readily prompted by the clinical features such as hyperphosphaturia, hypophosphatemia, low serum vitamin D3 levels, elevated serum fibroblast growth factor 23 levels, and osteomalacia. However, the causative tumor is frequently hidden in an unusual anatomical site and often goes undetected by conventional imaging, such as computed tomography (CT), while a permanent cure of the disease will only rely on exact localization and completely removal of the tumor.

Since mesenchymal tumors express somatostatin receptors (SSR), molecular imaging using radiolabeled somatostatin analogs may be one of the best ways to detect the small, occult tumors. 111In- and 99mTc-labeled octreotide and analogs have been proved useful to detect mesenchymal tumor and other SSR-positive tumors. However, the scintigraphy is insufficient to provide high-resolution images and precise anatomical information. In this study, a novel approach was proposed for exact localization of mesenchymal tumors through positron emission tomography (PET) imaging with 68Ga-DOTATATE and co-registration with CT. 68Ga-DOTATATE PET/CT is a novel method that might have improved sensitivity and resolution specifically for SSR-positive tumors, including the causative tumor of oncogenic osteomalacia.

The investigators will scan the patients in suspicion of oncogenic osteomalacia and the confirmed oncogenic osteomalacia patients in suspicion of relapse or with residual tumor after surgery, and compare it to 99mTc-HYNIC-TOC SPECT/CT and 18F-FDG PET/CT of the same patients. The aim of the study was to see if 68Ga-DOTATATE PET/CT can detect more tumors with higher resolution and more exact localization, and then help to develop optimal treatment strategy and improves patient care.

ELIGIBILITY:
Inclusion Criteria:

* In suspicion of oncogenic osteomalacia according to the clinical features such as hyperphosphaturia, hypophosphatemia, low serum vitamin D3 levels, and osteomalacia. Or prior oncogenic osteomalacia patients in suspicion of relapse or with residual tumor
* At least 18 years old
* Able to provide informed consent

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Renal function: serum creatinine >3.0 mg/dL (270 μM/L)
* Liver function: any hepatic enzyme level more than 5 times upper limit of normal.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Patients not able to enter the bore of the PET/CT scanner.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Any other medical condition that, in the opinion of the Investigator, may significantly interfere with study compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number and location of lesions detected by 68GA-DOTATATE PET/CT compared to 99mTc-HYNIC-TOC SPECT/CT and/or 18F-FDG PET/CT | 1 year
  Determine if the 68Ga-DOTATATE PET/CT changes care plans compared to conventional imaging/diagnostic techniques (99mTc-HYNIC-TOC SPECT/CT, and/or 18F-FDG PET/CT, MRI, CT, ultrasonography).

SECONDARY OUTCOMES:
Number of participants and kinds of adverse events as a measure of safety | One year
  Determine if any adverse effects are associated with the scan and the number of patients that experience them.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, MD, Study Chair — Department of Nuclear Medicine, Peking Union Medical College Hospital
Locations (1):
- Department of Nuclear Medicine, Peking Union Medical College Hopital, Beijing, China

IPD SHARING:
Plan to Share IPD: No